CLINICAL TRIAL: NCT05832970
Title: Brief Skin Cooling Induces Muscle Spindle Sensitivity With Heightened Sympathetic Outflow
Brief Title: Cooling Induces Motor Facilitation With Sympathetic Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ilhan KARACAN, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CIMFSA
Record Dates: First submitted 2023-04-03; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Cryotherapy Effect
Keywords: muscle spindle; sympathetic outflow; motor facilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hand cooling (Experimental): Records will be taken for Baseline electromyography, Heart rate, H-reflex, and T-reflex measurements before, during, and at 0, 3, 6, 9, 12, and 15. minutes before applying 2-4 degrees Celsius cold to the back of the hand in this group.
  Interventions: Other: Brief skin cooling

INTERVENTIONS:
Other: Brief skin cooling — Brief skin cooling will be applied to the hand using the cold-bath immersion

SUMMARY:
Cryotherapy has beneficial effects such as motor facilitation, increase isometric force generation, and reduce spasticity.

It is known that the muscle spindle has sympathetic innervation. Muscle spindle sensitivity increase with sympathetic activity. This research has three hypotheses: First, short-term cold application to the skin increases sympathetic activity. Second, there is an increase in muscle spindle sensitivity with increased sympathetic activity. Third, the effect of short-term cold on muscle spindle sensitivity continues until the skin temperature returns to normal. The purpose of this research is to test these hypotheses.

DETAILED DESCRIPTION:
Cryotherapy is a frequently used treatment method in sports medicine and rehabilitation due to its beneficial neuromuscular effects. Its main beneficial effects are motor facilitation, increase isometric force generation, and reduce spasticity. The motor effects of cryotherapy may differ depending on the duration of application, the coolant used agent (ice, ice water, coolant spray, etc.), and the thickness of the subcutaneous adipose tissue. The short-term cold application increases the force of contraction with motor facilitation. As the cold application period gets longer, the effects of the cold that inhibit motor functions such as gamma motor neuron inhibition, muscle spindle inhibition, and muscle conduction block come to the fore.

It is known that the muscle spindle has sympathetic innervation. It has been reported in recent studies that mental arithmetic, cold application to the skin, isometric contraction of remote muscles, and ischemia increase muscle spindle sensitivity through increased sympathetic activity. However, there are very limited studies showing that cold application increases muscle spindle sensitivity through increased sympathetic activity. On the other hand, in terms of determining treatment and rehabilitation strategies, it is important to know how long the effect of the cold application on muscle spindle sensitivity continues. However, it is not clear how long the effect of the cold application on muscle spindle sensitivity lasts after the cold application ends. There is a widespread belief that the motor facilitation effect of cryotherapy can occur with the stimulation of cutaneous cold receptors. Considering this view, it can be thought that the effect of the short-term cold application on muscle spindle sensitivity continues until the skin temperature returns to normal. This research has three hypotheses: First, short-term cold application to the skin increases sympathetic activity. Second, there is an increase in muscle spindle sensitivity with increased sympathetic activity. Third, the effect of short-term cold on muscle spindle sensitivity continues until the skin temperature returns to normal. The purpose of this research is to test these hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy
* Being a young adult (20-45 years old)
* Volunteer

Exclusion Criteria:

* Scar, dermatitis, etc. in the skin tissue where the superficial electromyography electrode will be placed
* Upper extremity bone and joint disease, history of neuromuscular disease
* Heart disease, Hypertension
* Cold intolerance

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2023-04-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Heart rate | Baseline (pre-cold pressor test) and 0, 3, 6, 9, 12, 15 minutes post-cold pressor test
  Heart rate will be monitored with DII derivation electrocardiographic recording.Heart rate will be reported as beats per minute.
Change from baseline in Soleus H-reflex | Baseline (pre-cold pressor test) and 0, 3, 6, 9, 12, 15 minutes post-cold pressor test
  By stimulating the tibial nerve with an electrical current, the Soleus H-reflex will be obtained. Its peak to peak amplitude will be measured in microvolts.
Change from baseline in T-reflex | Baseline (pre-cold pressor test) and 0, 3, 6, 9, 12, 15 minutes post-cold pressor test
  Soleus T-reflex will be obtained by hitting the Achilles tendon with the electronic reflex hammer. Its peak to peak amplitude will be measured in microvolts.

SECONDARY OUTCOMES:
Skin temperature | Baseline (pre-cold pressor test) and 0, 3, 6, 9, 12, 15 minutes post-cold pressor test
  The skin temperature of the back of the hand exposed to the cold application will be measured with an infrared thermometer and the results will be reported in degrees Celsius.

CONTACTS AND LOCATIONS:
Overall Officials: ILHAN KARACAN, MD, Prof, Principal Investigator — İstanbul Physical Therapy Rehabilitation Training & Research Hosptial
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training & Research Hospital, Istanbul, Turkey (Türkiye)